CLINICAL TRIAL: NCT04853940
Title: Respiratory Muscle Function, Dyspnea, Exercise Capacity and Quality of Life in Severe COVID19 Patients After ICU Discharge: a 6 Months Follow-up Observational Study
Brief Title: Respiratory Muscle Function, Dyspnea, Exercise Capacity and Quality of Life in Severe COVID19 Patients
Status: Completed | Type: Observational
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Maria Natividad Seisdedos Nunez, Senior Physiotherapist, MSc, Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal
Other Study IDs: 419/20
Record Dates: First submitted 2021-04-12; First posted 2021-04-22 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Covid19
Keywords: COVID19; Diaphragm ultrasound; Respiratory muscle strength; Dyspnea; Exercise Capacity; Quality of life; Post-ICU outcomes
MeSH Terms: conditions — COVID-19; Dyspnea | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Data collection and clinical testing of subjects — 6-months follow-up with clinical testing at 3 and 6 months

SUMMARY:
Further knowledge regarding sequelae in severe COVID-19 patients who have required ICU admission for invasive mechanical ventilation is still needed. Available evidence suggests ongoing respiratory impairment and impact in quality of life.

DETAILED DESCRIPTION:
PURPOSE: To evaluate post-ICU clinical outcomes in severe COVID-19 ICU survivors.

DESIGN: A prospective observational study conducted in public hospital in Madrid, Spain.

METHODS:

Participants: patients diagnosed with severe COVID-19 who have survived ICU admission for invasive mechanical ventilation and have been discharged from hospital.

Intervention: Patients will be invited to attend follow-up visits at the hospital for assessments 3 months and 6 months after ICU discharge.

Outcome measures: Tests of respiratory muscles function will include ultrasonography of the diaphragm muscle to measure diaphragm thickness (DT), diaphragm thickening ratio (TR) and diaphragm excursion (DE); respiratory muscle strength measurement to obtain Maximal Inspiratory Pressure (MIP), Maximal Expiratory Pressure (MEP) and Maximal Sniff Nasal Inspiratory Pressure (SNIP); functional exercise capacity will be assessed with the Six Minutes Walk Test (6MWT); dyspnea and health-related quality of life will be evaluated with the Modified Medical Research Council Scale (mMRC Scale) and the Saint George's Respiratory Questionnaire (SGRQ). Data on participants' demographics and clinical data will also be collected.

Statistical Analysis: Descriptive statistics will be used to summarise data. Spearman's correlation coefficients will be used to explore associations between variables.

CONCLUSIONS AND SIGNIFICANCE OF THE RESEARCH: Understanding post-ICU clinical outcomes in patients with severe COVID-19 may help develop future prevention, therapeutic and follow-up strategies that improve quality of care and outcomes

ELIGIBILITY:
Inclusion Criteria:

* ⋧18 years old,
* subjects diagnosed with COVID-19 confirmed by positive SARS-CoV-2 PCR testing who require admission to ICU for invasive mechanical ventilation
* invasive ventilation > 24 hours.

Exclusion Criteria:

* pre-existing cognitive impairment,
* communication/language barrier
* any concurrent physical or mental health condition/ impairment that prevents subjects from taking part in evaluations or providing informed consent
* loss of independent walking ability (with or without walking aids) prior to hospitalisation defined by a score of ≤2 on the mobility item of the modified Barthel Index,
* pregnancy,
* any injuries/surgery that requires medical bed rest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with COVID19 pneumonia who are discharged from the Ramón y Cajal University Hospital ICU from 1 October 2020 to 28 February 2021 will be eligible for the study
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure (MIP) (centimetres of water, cmH20) | < 3 months after ICU discharge
  It is the greater pressure which may be generated during maximal inspiration by the inspiratory muscles.
Maximal Inspiratory Pressure (MIP) (centimetres of water, cmH20) | within 6 months after ICU discharge
  It is the greater pressure which may be generated during maximal inspiration by the inspiratory muscles.

SECONDARY OUTCOMES:
Diaphragm Thickening Ratio during deep breathing (centimetres) | within 3 months after ICU discharge
  B-mode Diaphragm ultrasound will be performed to measure diaphragm thickening ratio during deep breathing. Diaphragm Thickening Ratio = Diaphragm Thickness at Functional Residual Capacity/ Diaphragm thickness at Total Lung Capacity.
Diaphragm Thickening Ratio during deep breathing (centimetres) | within 6 months after ICU discharge
  B-mode Diaphragm ultrasound will be performed to measure diaphragm thickening ratio during deep breathing. Diaphragm Thickening Ratio = Diaphragm Thickness at Functional Residual Capacity/ Diaphragm thickness at Total Lung Capacity.
Diaphragm Thickening Ratio during quiet breathing (centimetres) | within 3 months after ICU discharge
  B-mode Diaphragm ultrasound will be performed to measure diaphragm thickening ratio at Tidal Volume. Diaphragm Thickening Ratio = Diaphragm Thickness at the end of a quiet expiration/ Diaphragm thickness at the end of a quiet inspiration.
Diaphragm Thickening Ratio during quiet breathing (centimetres) | within 6 months after ICU discharge
  B-mode Diaphragm ultrasound will be performed to measure diaphragm thickening ratio at Tidal Volume. Diaphragm Thickening Ratio = Diaphragm Thickness at the end of a quiet expiration/ Diaphragm thickness at the end of a quiet inspiration.
Diaphragm Excursion during deep breathing (centimetres) | within 3 months after ICU discharge
  M-mode Diaphragm Ultrasound imaging will be performed to measure diaphragm excursion during deep breathing defined as the displacement (centimetres) of the diaphragm between Functional Residual Capacity and Total Lung Capacity
Diaphragm Excursion during deep breathing (centimetres) | within 6 months after ICU discharge
  M-mode Diaphragm Ultrasound imaging will be performed to measure diaphragm excursion during deep breathing defined as the displacement (centimetres) of the diaphragm between Functional Residual Capacity and Total Lung Capacity.
Maximal Expiratory Pressure (MEP) (cmH20) | within 3 months after ICU discharge
  It is the greater pressure which may be generated during maximal expiration by the inspiratory muscles.
Maximal Expiratory Pressure (MEP) (cmH20) | within 6 months after ICU discharge
  It is the greater pressure which may be generated during maximal expiration by the inspiratory muscles.
Modified Medical Research Council (mMRC) Dyspnea score | within 3 months following ICU discharge
  Dyspnea will be measured with the mMRC Dyspnea scale (range: 0-4, higher values indicating higher level of dyspnea)
Modified Medical Research Council (mMRC) Dyspnea score | within 6 months following ICU discharge
  Dyspnea will be measured with the mMRC Dyspnea scale (range: 0-4, higher values indicating higher level of dyspnea)
6-Minutes Walk Test (6MWT) (metres) | within 3 months following ICU discharge
  The 6MWT will be used to measure exercise capacity
6-Minutes Walk Test (6MWT) (metres) | within 6 months following ICU discharge
  The 6MWT will be used to measure exercise capacity
Saint George's Respiratory Questionnaire (SGRQ) score | within 3 months following ICU dischargemonths following ICU discharge
  The SGRQ is used to measure health-related quality of life (range: 0-100, higher scores represent higher impairment in quality of life)
Saint George's Respiratory Questionnaire (SGRQ) score | within 6 months following ICU dischargemonths following ICU discharge
  The SGRQ is used to measure health-related quality of life (range: 0-100, higher scores represent higher impairment in quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Luís López-González, BSc,MSc, Principal Investigator — Fundación Ramón y Cajal
Locations (1):
- ICU. Ramón y Cajal University Hospital, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided